CLINICAL TRIAL: NCT05195632
Title: Multicenter, Open-label, Phase II Study With a Safety Lead-in Part Investigating the Efficacy, Safety and Pharmacokinetics of Encorafenib and Binimetinib Combination in BRAF V600E Mutated Chinese Patients With Metastatic Non-Small Cell Lung Cancer Who Are BRAF- and MEK Inhibitor Treatment-naïve
Brief Title: Phase II Study Investigating the Combination of Encorafenib and Binimetinib in BRAF V600E Mutated Chinese Patients With Metastatic Non-Small Cell Lung Cancer
Acronym: OCEANII
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W00090GE203; CTR20212962 (Registry Identifier: Center for Drug Evaluation (CDE)); CTR20212961 (Registry Identifier: Center for Drug Evaluation (CDE))
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Encorafenib; Binimetinib; Lung Cancer; BRAF-inhibitor; MEK-inhibitor; BRAF V600E -mutated Chinese patients; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — encorafenib; binimetinib

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, phase 2 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Safety Lead-in and Pivotal arm) (Experimental): Encorafenib will be administered as a fixed, flat oral dose of 450 mg QD in combination with binimetinib as a fixed, flat oral dose of 45 mg BID.
  Interventions: Drug: Encorafenib; Drug: Binimetinib

INTERVENTIONS:
Drug: Encorafenib — Hard capsule
  Other Names: PF-07263896 or W0090 (in Europe), LGX818 (in US), ONO-7702 (in Japan)
Drug: Binimetinib — Film-coated tablet
  Other Names: W0074 (in Europe), MEK162 (in US), ARRY-438162 (in US), ONO-7703 (in Japan)

SUMMARY:
This is a phase 2, multicenter, single-arm study with a safety lead-in to investigate the efficacy, safety and pharmacokinetics of encorafenib 450 mg once daily (QD) in combination with binimetinib 45 mg twice daily (BID) (Combo450) in adult Chinese participants with metastatic unresectable stage IV BRAF V600E mutant NSCLC, who are BRAF- and MEK-inhibitor treatment-naïve and are either previously untreated or have had one line of prior therapy in metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

If a participant has a BRAF V600E mutational status confirmed as per local assessment, the participant might enter the main screening directly.

All the following inclusion criteria must be met for a participant to be eligible to be included in this study:

1. Provide a signed and dated screening Informed Consent Form (ICF).
2. Chinese male or female with age ≥ 18 years old for China mainland and ≥ 20 years old for Taiwan at the time of the screening informed consent.
3. Documented histology- and/or cytology-confirmed metastatic unresectable Non-small cell lung cancer (NSCLC (i.e. Adenocarcinoma (ADC), large cell carcinoma, squamous cell carcinoma (SCC)).
4. Presence of B-Raf Proto-Oncogene, Serine/Threonine Kinase (BRAF) V600E mutation in tumor tissue previously determined by a local assay at any time prior to screening or by the central laboratory.
5. Able to provide a sufficient amount of representative tumor specimen (primary or metastatic, archived or newly obtained) for central prospective laboratory testing of BRAF mutation status and comparison of central BRAF V600E testing in the clinical study to BRAF V600E testing with a candidate companion diagnostic.
6. BRAF- and Mitogen-activated protein kinase kinase (MEK)-inhibitor treatment-naïve participants and previously untreated or have had one line of prior therapy in metastatic setting.
7. At least one measurable disease as per investigator assessment, as defined by RECIST v1.1, which has neither been irradiated nor biopsied during the screening period.
8. Life expectancy ≥ 3 months.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
10. Adequate hematologic function at screening and baseline.
11. Adequate hepatic function at screening and baseline.
12. Adequate renal function at screening and baseline.
13. Able to comply with the study protocol as per investigator assessment including oral drug intake, complying scheduled visits, treatment plan, laboratory tests and other study procedures.
14. Women are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks, or child-bearing potential women must agree to take appropriate precautions to avoid pregnancy.
15. Men must agree not to father child until 90 days after the last dose of the study treatment.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible to be included in this study:

1. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs (encorafenib and binimetinib), or their excipients.
2. Documented Anaplastic lymphoma kinase (ALK) fusion oncogene, Reactive oxygen species (ROS) rearrangement or Epidermal growth factor receptor (EGFR) sensitizing or driver mutation.
3. Participants who have received more than one prior line of systemic therapy.
4. Receipt of anti-cancer medications or investigational drugs within the specified intervals before the first administration of study treatment.
5. Symptomatic brain metastases or other active Central nervous system (CNS) metastases.
6. Leptomeningeal disease.
7. Participant has not recovered to ≤ Grade 1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting study treatment.
8. Current use of prohibited medication ≤ 1 week prior to start of the study treatment and/or concomitantly.
9. Impairment of gastrointestinal function or disease which may significantly alter the absorption of oral study treatment.
10. Impaired cardiovascular function or clinically significant cardiovascular diseases
11. History of thromboembolic or cerebrovascular events within 3 months prior to starting the study treatments
12. History or evidence of retinal pathology considered as risk factor for Retinal vein occlusion (RVO) or neovascular macular degeneration.
13. Concurrent neuromuscular disorder associated with the potential of elevated Creatine phosphokinase (CPK)
14. Participants with active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) or any other severe viral active infection (e.g. SARS-CoV-2 infection)
15. Evidence of active, non-infectious pneumonitis, history of interstitial lung disease that required oral or intravenous glucocorticosteroids for management.
16. Known history of a positive test for Human immunodeficiency virus (HIV) or known Acquired Immunodeficiency Syndrome (AIDS). Testing for HIV must be performed at sites where mandated locally.
17. Participants who have had major surgery (e.g. inpatient procedure with regional or general anesthesia) within 6 weeks prior to start of study treatment.
18. Participants with concurrent or history of another malignancy within 2 years of study entry Except:

    1. Bowen's disease
    2. Cured basal cell or cutaneous squamous cell carcinoma (CuSCC)
    3. Gleason 6 prostate cancer
    4. Treated in-situ carcinoma of cervix
19. Participant's conditions that contraindicates the use of study treatments and may affect interpretation of results or may render the participant at high risk from treatment complications.
20. Pregnant (confirmed by positive serum beta-human chorionic gonadotropin (ß-HCG) test), lactating or breast-feeding women.
21. Is a family member of the investigator or any associate, colleague, and employee assisting in the conduct of the study (secretary, nurse, technician).
22. Is in a position likely to represent a conflict of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-In (SLI) Part: Incidence of Dose-limiting toxicities (DLTs) | Cycle 1; Each cycle is 28 days
  Incidence of DLTs experienced during the Cycle 1 (days 1 to 28) after the first dose of study treatment. DLT rate defined as the number of DLT-evaluable participants with DLTs in the first 28 days after first dose of study treatment in the SLI (DLT-evaluation period), divided by the number of DLT-evaluable participants.
Pivotal Part: Confirmed objective response rate (cORR) | Cycle 1 Day 1 through safety follow-up visit (30 days after end of treatment (EOT) visit or 7 days after EOT visit/last dose if EOT not performed), approximately up to 18 months. Each cycle is 28 days.
  cORR defined as the percentage of participants who have achieved a complete response (CR) or partial response (PR) as determined by Independent Central Review (ICR) of radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Proportion of patients who have achieved a confirmed Best Overall Response (cBOR) of CR or PR as determined by per RECIST v1.1 and corresponding exact two-sided binomial 95% Confidence interval (CI).

SECONDARY OUTCOMES:
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of encorafenib: Area under the curve (AUC) | Cycle 1 Day 1; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of encorafenib: Minimum serum concentration (Cmin) | Cycle 1 Day 1; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of encorafenib: Maximum serum concentration (Cmax) | Cycle 1 Day 1; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of binimetinib: Area under the curve (AUC) | Cycle 1 Day 1; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of binimetinib: Minimum serum concentration (Cmin) | Cycle 1 Day 1; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of binimetinib: Maximum serum concentration (Cmax) | Cycle 1 Day 1; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of encorafenib metabolite (LHY746): Area under the curve (AUC) | Cycle 1 Day 1; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of encorafenib metabolite (LHY746): Minimum serum concentration (Cmin) | Cycle 1 Day 1; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of encorafenib metabolite (LHY746): Maximum serum concentration (Cmax) | Cycle 1 Day 1; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of binimetinib metabolite (AR00426032): Area under the curve (AUC) | Cycle 1 Day 1; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of binimetinib metabolite (AR00426032): Minimum serum concentration (Cmin) | Cycle 1 Day 1; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Safety Lead-In (SLI) Part: Pharmacokinetic (PK) parameter of binimetinib metabolite (AR00426032): Maximum serum concentration (Cmax) | Cycle 1 Day 1; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Safety Lead-In (SLI) Part: Incidence, nature and severity of treatment emergent adverse events (TEAEs) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Incidence, nature and severity of TEAEs graded as per NCI CTCAE v4.03, TEAEs leading to dose interruption, reduction and discontinuation, Treatment-emergent serious adverse events (SAEs), TEAEs leading to death.
Safety Lead-In (SLI) Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline clinical laboratory parameter: Hematology | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Hemoglobin, hematocrit, Red Blood Cells (RBC), White Blood Cells (WBC) with differential (absolutes values), platelet counts, neutrophils, lymphocytes, monocytes, basophils and eosinophils
Safety Lead-In (SLI) Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline clinical laboratory parameter: Chemistry | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Albumin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin and direct bilirubin, gamma glutamyl transferase (GGT), urea or blood urea nitrogen (BUN), creatinine, sodium, potassium, calcium, phosphate, chloride, uric acid, magnesium, Creatinine kinase (CK) (if total CK ≥ 3X upper limit of normal (ULN), then measure isoenzymes including Creatine Kinase BB, Creatine Kinase MB, Creatine Kinase MM), serum creatinine and myoglobin in blood and urinalysis test weekly; if there is no local capability to measure CK isoenzymes, then participants must be referred to a local hospital for appropriate management while central laboratory results are awaited. If a diagnosis of rhabdomyolysis is confirmed, then sites should liaise with their local hospitals regarding management of the participants and administration of study medication), total protein, glucose, lactate dehydrogenase (LDH), lipase and amylase.
Safety Lead-In (SLI) Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline clinical laboratory parameter: Coagulation | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Prothrombin time (PT), international normalized ratio (INR) and activated partial thromboplastin time (aPTT)
Safety Lead-In (SLI) Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline of dipstick urinalysis | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Dipstick measurements for specific gravity, pH, protein, glucose, bilirubin, ketones, leukocytes, and blood will be performed. Any clinically significant findings on dipstick will be followed up with a microscopic evaluation.
Safety Lead-In (SLI) Part: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes in vital signs from baseline of vital sign examinations. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Clinically notable elevated values: Systolic blood pressure (BP): ≥ 160 mmHg and an increase ≥ 20 mmHg from baseline; Diastolic BP: ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline; Heart rate: ≥ 120 beats/min (bpm) with increase from baseline of ≥ 15 bpm; Weight (kg) increase from baseline of ≥ 10%; Body temperature [°C] ≥ 37.5°C). Clinically notable low values: Systolic BP: ≤ 90 mmHg with decrease from baseline of ≥ 20 mmHg; Diastolic BP: ≤ 50 mmHg with decrease from baseline of ≥ 15 mmHg; Heart rate: ≤ 50 bpm with decrease from baseline of ≥ 15 bpm; Weight: ≥ 20% decrease from baseline; Body temperature [°C]: ≤ 36 °C. Number of participants with TEAEs related to notable changes to the vital signs after the start of study drug will be reported.
Safety Lead-In (SLI) Part: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of 12-lead electrocardiograms (ECGs) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  12-lead ECGs will be obtained using an internationally recognized 12-lead cardiograph. Clinically notable ECG values: QT [millisecond (ms)] and QT interval (ms) corrected for heart rate using Fridericia's formula (QTcF) intervals (ms): increase from baseline > 30 ms; increase from baseline > 60 ms, new > 450 ms, new > 480 ms, new > 500 ms. Heart rate (beats/min): increase from baseline > 25% to a value > 100 bpm, decrease from baseline > 25% and to a value < 50 bpm. Number of participants with TEAEs related to abnormal or notable changes to ECG parameters after the start of study drug will be reported.
Safety Lead-In (SLI) Part: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of echocardiogram or multigated acquisition (ECHO/MUGA) scans. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  ECHO/MUGA scan assess Left Ventricular Ejection Fraction (LVEF). Changes from baseline of LVEF measurements over time will be reported.
Pivotal Part: Confirmed Objective Response Rate (cORR) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  cORR as determined by investigator review of the radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Pivotal Part: Objective Response Rate (ORR) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  ORR as determined by investigator review and independent central review (ICR) of the radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Pivotal Part: Duration of Response (DOR) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  DOR defined as the time from first documented response (i.e. complete response (CR) or partial response (PR)) to the earliest documented disease progression, as determined by investigator review and independent central review (ICR) of radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death from any cause, whichever occurs first.
Pivotal Part: Disease Control Rate (DCR) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  DCR defined as the proportion of participants who have achieved a best overall response of complete response (CR), partial response (PR) or stable disease (SD) as determined by investigator review and independent central review (ICR) of radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Pivotal Part: Time to Progression (TTP) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  TTP defined as the time from first study treatment dose to the earliest documented disease progression as per investigator review and independent central review (ICR) of radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Pivotal Part: Progression Free Survival (PFS) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  PFS defined as the time from first study treatment dose to the earliest documented disease progression as per investigator review and independent central review (ICR) of radiographic disease assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurs first.
Pivotal Part: Overall Survival (OS) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  OS defined as the time from first study treatment dose to the date of death due to any cause.
Pivotal Part: Incidence, nature and severity of treatment emergent adverse events (TEAEs) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Incidence, nature and severity of treatment emergent adverse events (TEAEs) graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Pivotal Part: Treatment emergent adverse events (TEAEs) leading to dose interruption, reduction and discontinuation. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Incidence, nature and severity of TEAEs leading to dose interruption, reduction and discontinuation will be reported.
Pivotal Part: Incidence of treatment emergent serious adverse events (SAEs) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Incidence, nature and severity of SAE will be recorded and graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Pivotal Part: Incidence of treatment emergent adverse events (TEAEs) leading to death | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  TEAEs leading to deaths will be reported.
Pivotal Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline clinical laboratory parameter: Hematology | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Hemoglobin, hematocrit, Red Blood Cells (RBC), White Blood Cells (WBC) with differential (absolutes values), platelet counts, neutrophils, lymphocytes, monocytes, basophil and eosinophils
Pivotal Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline clinical laboratory parameter: Chemistry | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Albumin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin and direct bilirubin, gamma glutamyl transferase (GGT), urea or blood urea nitrogen (BUN), creatinine, sodium, potassium, calcium, phosphate, chloride, uric acid, magnesium, Creatinine kinase (CK) (if total CK ≥ 3X upper limit of normal (ULN), then measure isoenzymes (including all fractions), serum creatinine and myoglobin in blood and urinalysis test weekly; if there is no local capability to measure CK isoenzymes, then subjects must be referred to a local hospital for appropriate management while central laboratory results are awaited. If a diagnosis of rhabdomyolysis is confirmed, then sites should liaise with their local hospitals regarding management of the subjects and administration of study medication), total protein, glucose, lactate dehydrogenase (LDH), lipase and amylase.
Pivotal Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline clinical laboratory parameter: Coagulation | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Prothrombin time (PT), international normalized ratio (INR) and activated partial thromboplastin time (aPTT)
Pivotal Part: Incidence of treatment emergent adverse events (TEAEs) related to notable change from baseline of dipstick urinalysis. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Dipstick measurements for specific gravity, pH, protein, glucose, bilirubin, ketones, leukocytes, and blood will be performed. Any clinically significant findings on dipstick will be followed up with a microscopic evaluation.
Pivotal Part: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes in vital signs from baseline of vital sign examinations. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Clinically notable elevated values: Systolic blood pressure (BP): ≥ 160 mmHg and an increase ≥ 20 mmHg from baseline; Diastolic BP: ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline; Heart rate: ≥ 120 beats/min (bpm) with increase from baseline of ≥ 15 bpm; Weight (kg) increase from baseline of ≥ 10%; Body temperature [°C] ≥ 37.5°C). Clinically notable low values: Systolic BP: ≤ 90 mmHg with decrease from baseline of ≥ 20 mmHg; Diastolic BP: ≤ 50 mmHg with decrease from baseline of ≥ 15 mmHg; Heart rate: ≤ 50 bpm with decrease from baseline of ≥ 15 bpm; Weight: ≥ 20% decrease from baseline; Body temperature [°C]: ≤ 36 °C. Number of participants with TEAEs related to notable changes to the vital signs after the start of study drug will be reported.
Pivotal Part: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of 12-lead electrocardiograms (ECGs) | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  12-lead ECGs will be obtained using an internationally recognized 12-lead cardiograph. Clinically notable ECG values: QT [millisecond (ms)] and QT interval (ms) corrected for heart rate using Fridericia's formula (QTcF) intervals (ms): increase from baseline > 30 ms; increase from baseline > 60 ms, new > 450 ms, new > 480 ms, new > 500 ms. Heart rate (beats/min): increase from baseline > 25% to a value > 100 bpm, decrease from baseline > 25% and to a value < 50 bpm. Number of participants with TEAEs related to abnormal or notable changes to ECG parameters after the start of study drug will be reported.
Pivotal Part: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of echocardiogram or multigated acquisition (ECHO/MUGA) scans. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  ECHO/MUGA scan assess Left Ventricular Ejection Fraction (LVEF). Changes from baseline of LVEF measurements over time will be reported.
Pivotal Part: Incidence of targeted treatment emergent adverse events (TEAEs) of special interest. | Cycle 1 Day 1 through safety follow-up visit (30 days (+/- 3 days)) after last study treatment dose or before the initiation of subsequent anticancer therapy, whichever occurs first, approximately up to 18 months. Each cycle is 28 days.
  Number and percentage of participants with at least one event of adverse event (AE) of special interest (AESI) will be reported.
Pivotal Part: Pharmacokinetic (PK) parameter of encorafenib: Area under the curve (AUC) | Cycle 1 Day 1 and Cycle 2 Day 1 at pre-dose, and 1, 2, 4, 6 hours post-dose; Cycle 1 to Cycle 6 at pre-dose for sparse samples; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of encorafenib: Minimum serum concentration (Cmin) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of encorafenib: Maximum serum concentration (Cmax) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of binimetinib: Area under the curve (AUC) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of binimetinib: Minimum serum concentration (Cmin) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of binimetinib: Maximum serum concentration (Cmax) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of encorafenib metabolite (LHY746): Area under the curve (AUC) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of encorafenib metabolite (LHY746): Minimum serum concentration (Cmin) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of encorafenib metabolite (LHY746): Maximum serum concentration (Cmax) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of binimetinib metabolite (AR00426032): Area under the curve (AUC) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Area under the curve (AUC) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of binimetinib metabolite (AR00426032): Minimum serum concentration (Cmin) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Minimum serum concentration (Cmin) will be calculated and reported.
Pivotal Part: Pharmacokinetic (PK) parameter of binimetinib metabolite (AR00426032): Maximum serum concentration (Cmax) | Cycle 1 Day 1 and Cycle 2 Day 1; Cycle 1 to Cycle 6 at pre-dose; Each cycle is 28 days
  Maximum serum concentration (Cmax) will be calculated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen Univ. Cancer Center
Locations (34):
- China (33):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The Second Hospital of Dalian University, Dalian
  - Fujian Medical University Union Hospital, Fuzhou
  - Fuzhou Tuberculosis Prevention and Control Hospital of Fujian Province (Fuzhou Pulmonary Hospital of Fujian), Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Hainan General Hospital, Haikou
  - First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Zhejiang University School of Medicine, Sir Run Run Shaw Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Union Hospital Tongji medical college Huazhong University of Science and Technology, Wuhan
  - The Northern Jiangsu People's Hospital, Yangzhou
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No